CLINICAL TRIAL: NCT05876767
Title: A Randomized, Double-blind, Placebo-controlled Study of the Tolerability, Pharmacokinetics and Pharmacodynamics of Ascending Single and Repeated Subcutaneous Doses of SAR444336 in Healthy Adult Participants
Brief Title: Tolerability, Pharmacokinetics and Pharmacodynamics of Ascending Single and Repeated Doses of SAR444336 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TDU17072-TDR17161
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAR444336 (Experimental): SAR444336
  Interventions: Drug: SAR444336
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR444336 — Single or repeated dose subcutaneous injection
  Arms: SAR444336
Drug: Placebo — Single or repeated dose subcutaneous injection
  Arms: Placebo

SUMMARY:
This phase 1 study will assess the safety and tolerability, and characterize the pharmacokinetic (PK) and pharmacodynamic (PD) profile of SAR444336 in healthy subjects following single- and repeated-dose administrations as a first step in clinical development prior to administering this new investigational medicinal product (IMP) to patients.

DETAILED DESCRIPTION:
The anticipated study duration per participant is up to 10 weeks in Part 1.

* Screening: 2 to 28 days prior to dosing (Day -28 to Day -2)
* Treatment period: Day -1 to Day 29 post dose including
* Institutionalization: Day -1 until Day 8
* Ambulant period including repeat PK and PD blood sampling and ambulant visits: Day 9 to Day 29
* Follow-up period: Day 30 to Day 43

The anticipated study duration per participant is up to 17 weeks in Part 2.

* Screening: 2 to 28 days prior to dosing (Day -28 to Day -2)
* Treatment period: Day -1 to Day 57 (Q2W/3 doses or Q4W/2 doses) or Day -1 to Day 85 (Q4W/3 doses), or Day -1 to Day 50 (Q3W) including
* Institutionalization: Day -1 until Day 3
* Ambulant period including repeat PK and PD blood sampling, ambulant visits and 24 hours institutionalization after 2nd and/or 3rd dose: Day 4 to Day 57 (Q2W/3 doses, Q4W/2 doses), Day 4 to Day 85 (Q4W/3 doses) or Day 50 (Q3W)
* Follow-up period: Day 58 to Day 71 (Q2W/3 doses or Q4W/2 doses), Day 71 to Day 85 (Q4W/3 doses) or Day 51 to Day 64 (Q3W)

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between 18 and 55 years of age inclusive.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECG.
* Laboratory values within normal range unless the abnormality is considered not clinical relevant by the investigator. The following parameters, however, must be within normal range: platelet count, and CRP. ALT, AST, total bilirubin (unless the participant has documented or suspected Gilbert syndrome) should be <1.25 ULN and serum creatinine should be < ULN.
* Eosinophils <500 cells/µL
* Normal vital signs after 10 minutes resting in supine position
* Standard 12-lead ECG parameters after 10 minutes resting in supine position in the normal ranges and normal ECG tracing unless the Investigator considers an ECG tracing abnormality to be not clinically relevant.
* Body weight between 50 - 110 kg (inclusive) and body mass index (BMI) between 18 - 30 kg/m2 (inclusive) at screening.
* Only for part 2: Fitzpatrick skin type I - III

Exclusion Criteria:

* Any disease associated with immune system dysfunction.
* Known polyethylene glycol allergy
* Only for Part 2: Known seafood allergy
* Any current active viral, bacterial or fungal infection or any medically relevant infection having occurred within 3 weeks before inclusion.
* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, autoimmune, systemic, ocular, or infectious disease, or signs of acute illness that would pose an unacceptable risk to the subject in the opinion of the investigator.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only, more than twice a month).
* Blood donation >500 mL within 2 months before inclusion.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥30 mmHg within 3 minutes when changing from supine to standing position.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician, except for history of mild allergic diseases which are not active at the time of inclusion and considered not clinically relevant in the opinion of the investigator.
* History or presence of drug or alcohol abuse.
* Smoking regularly more than 10 cigarettes or equivalent per week, unable to stop smoking during the study (occasional smoker can be enrolled).
* Excessive consumption of beverages containing xanthine bases.
* Presence or history of any atopic disease.
* for Part 1: Non-live booster COVID-19 vaccination within 14 days before randomization. First (and second, if applicable) COVID-19 vaccinations are not allowed within 4 weeks before randomization.
* for Part 2: Non-live vaccines including Covid-19: last administration of a vaccine within 4 weeks before randomization.
* Live vaccines: Last administration of a vaccine within 3 months before randomization; Immunomodulatory medication within 60 days before screening.
* Only for Part 2: Participants with known previous exposure to KLH.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication; any vaccination within the last 28 days (except COVID-19 booster vaccination) and any biologics (antibody or its derivatives) given within 4 months before inclusion.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, antihepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-HIV1 and anti HIV2 Ab.
* Positive result on urine drug screen.
* Positive alcohol breath test.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of subjects with treatment-emergent adverse events (TEAEs) | Until Day 43
  Clinical laboratory evaluations including eosinophils, procalcitonin, and c-reactive protein (CRP), Vital signs, 12-lead electrocardiogram (ECG)
Part 2: Number of subjects with treatment-emergent adverse events (TEAEs) | Until Day 85
  Clinical laboratory evaluations including eosinophils, procalcitonin, and c-reactive protein (CRP), Vital signs, 12-lead electrocardiogram (ECG)

SECONDARY OUTCOMES:
Plasma PK parameters: Cmax | Until Day 29 and Day 85
  Maximum plasma concentration observed
Plasma PK parameters: tmax | Until Day 29 and Day 85
  Time to reach Cmax
Plasma PK parameters: AUClast | Until Day 29 and Day 85
  Area under the plasma concentration versus time curve over the dosing interval from time 0 until the last concentration above the limit of quantification
Plasma PK parameters: AUC | Until Day 29 and Day 85
  Area under the plasma concentration versus time curve extrapolated to infinity
Plasma PK parameters: t1/2z | Until Day 29 and Day 85
  Terminal half-life
Plasma PK parameters: CL/F | Until Day 29 and Day 85
  Apparent total body clearance after a single extravascular dose
Anti-SAR444336 antibodies | Until Day 29 and Day 85

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Investigational Site Number :5280001, Leiden, Leiden
  - Investigational Site Number :5280002, Groningen, Provincie Groningen

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TDU17072 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25471&tenant=MT_SNY_9011
- See also: TDR17161 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25455&tenant=MT_SNY_9011